CLINICAL TRIAL: NCT02005315
Title: A Phase 1b Dose Escalation Study of Vantictumab (OMP-18R5) in Combination With Nab-Paclitaxel and Gemcitabine in Patients With Previously Untreated Stage IV Pancreatic Cancer
Brief Title: A Study of Vantictumab (OMP-18R5) in Combination With Nab-Paclitaxel and Gemcitabine in Previously Untreated Stage IV Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18R5-003
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Cancer; Stage IV Pancreatic Cancer
Keywords: Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vanctictumab (OMP-18R5) (Experimental): Vantictumab will be administered by intravenous (IV) infusion.
  Interventions: Drug: Vantictumab; Drug: Nab-Paclitaxel; Drug: Gemcitabine
- Nab-Paclitaxel (Experimental): Nab-Paclitaxel will be administered by intravenous (IV) infusion.
  Interventions: Drug: Vantictumab; Drug: Nab-Paclitaxel; Drug: Gemcitabine
- Gemcitabine (Experimental): Gemcitabine will be administered by intravenous (IV) infusion.
  Interventions: Drug: Vantictumab; Drug: Nab-Paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Vantictumab — Administered intravenous (IV) infusion.
  Other Names: OMP-18R5
Drug: Nab-Paclitaxel — Nab-Paclitaxel will be administered by intravenous (IV) infusion.
Drug: Gemcitabine — Gemcitabine will be administered by intravenous (IV) infusion.

SUMMARY:
This is an open-label Phase 1b dose-escalation study to assess the safety, tolerability, and PK of vantictumab when combined with nab-paclitaxel and gemcitabine.

DETAILED DESCRIPTION:
Once the maximum tolerated dose (MTD) or maximum administered dose (MAD) has been determined, up to 10 patients may be enrolled in the cohort-expansion phase to better characterize the safety, tolerability and PK of vantictumab combined with nab-paclitaxel and gemcitabine. Up to approximately 34 patients may be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥18 years
* Histologically documented Stage IV ductal adenocarcinoma of the pancreas
* Availability of tumor tissue, either archival FFPE or obtained at study entry through fresh biopsy
* ECOG performance status of 0 or 1
* Adequate hematologic and end-organ function
* Evaluable or measurable disease per RECIST v1.1
* For women of childbearing potential and men with partners of childbearing potential, agreement to use two effective forms of contraception

Exclusion Criteria:

* Prior therapy before Day 1 of Cycle 1 for the treatment of Stage IV pancreatic cancer
* Prior adjuvant therapy for the treatment of ductal adenocarcinoma of the pancreas
* Known hypersensitivity to any component of study treatments
* Known brain metastases, uncontrolled seizure disorder, or active neurologic disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Phase 1b: Safety and tolerability of vantictumab in combination with nab-paclitaxel and gemcitabine in patients with previously untreated Stage IV pancreatic cancer | Subjects will be treated and observed for DLT through the end of the first cycle (Days 0-28)
  The maximum tolerated dose (MTD) will be determined in patients treated with vantictumab in combination with weekly nab-paclitaxel

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of vantictumab when administered in combination with nab-paclitaxel and gemcitabine to patients with previously untreated Stage IV pancreatic cancer | Vantictumab will be administered IV on Days 1 and 15 of each 28-day cycle. Nab-paclitaxel and gemcitabine will be administered IV on Days 1, 8, and 15 of each cycle.
  Apparent half life, AUC, clearance, volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Romnee Clark, MD, Principal Investigator — Indiana University Institutional Review Board (IRB)
Locations (5):
- United States (5):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Hospital Anschutz Cancer Pavillion, Aurora, Colorado
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee